CLINICAL TRIAL: NCT02506413
Title: Replicating MamaToto in Rural Tanzania
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Catholic University of Health and Allied Sciences (Other)
Responsible Party: Principal Investigator, Jennifer L. Brenner, Dr. Jennifer L. Brenner, University of Calgary
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IRT #39
Record Dates: First submitted 2015-07-01; First posted 2015-07-23 (Estimated); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Maternal Death; Newborn Death
Keywords: Maternal and Newborn Health
MeSH Terms: conditions — Maternal Death; Perinatal Death

STUDY DESIGN:
Intervention Model Description: This study was part of a longitudinal implementation evaluation using an effectiveness-intervention hybrid (Type 2) design and a RE-AIM evaluation model.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MNCH Intervention Package (Other): The division assigned to this arm received a comprehensive Maternal and Newborn Health (MNH) intervention package using the 'MamaToto Process'. Key intervention activities included:
  1. engaging district leaders in district health system strengthening;
  2. strengthening health facility-based MNH services; and
  3. establishing a Maternal, Newborn, and Child Health focused lay Community Health Worker program.
  Interventions: Other: MamaToto Package

INTERVENTIONS:
Other: MamaToto Package — The MamaToto Package (later called "Mama na Mtoto" for the Tanzanian context) was an MNCH intervention built upon prior successes in Uganda and adapted to meet the needs in Misungwi District in Tanzania. The intervention included low-cost programming that built upon the existing district health system structure and resources in order to strengthen the MNH capacity and training of the district, health facilities, and community health workers.
  Other Names: Mama na Mtoto

SUMMARY:
This study aimed to adapt and implement a district-led, policy-based, low cost Maternal and Newborn Health (MNH) intervention package using the MamaToto process, proven successful in Uganda, in rural Tanzania. The investigators hypothesized that the 'MamaToto Package' will be successfully implemented in the Misungwi District and will be effective in improving key maternal and newborn health indicators of study participants.

DETAILED DESCRIPTION:
This study collected baseline data on indicators related to pre-natal care, delivery, post-natal care, treatment of childhood illnesses and family planning. Data collection tools/strategies included 1) a mapping exercise, 2) health facility audit 3) household surveys and 4) exit interviews. Data was collected at baseline and endline. Operational data was collected throughout the life of the study. Results were used to inform implementation of interventions that aim to improve health facility capacity to deliver good quality care to women and children and to strengthen families and communities to better advocate for and engage in activities that promote healthier women and children.

Mapping data was collected in two districts 1) Misungwi and 2) Kwimba. Baseline and endline data was collected in Misungwi only. The intervention began in Misungwi in Years 1 and 2 and then rolled out to Kwimba in Year 3.

ELIGIBILITY:
Inclusion Criteria:

* Randomly selected households (30) living in selected hamlets with a competent participant of greater than 15 years of age
* All women of reproductive age (age 15-49 years old) living in selected households in selected hamlets

Exclusion Criteria:

* Households with participants that are away for an extended time or have no one home at the time of survey completion

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 8323 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Proportion of live births attended by a skilled health provider | Change between pre (baseline) and post (endline-up to 36 months) intervention
  Percentage of women (15-49 year old) with at least one recent live birth (past two years) reporting their last delivery being attended to by a skilled health personnel (doctor, nurse, midwife, clinical officer or auxiliary midwife)

SECONDARY OUTCOMES:
Proportion of women receiving postnatal care <48H | Change between pre (baseline) and post (endline-up to 36 months) intervention
  Percentage of women (15-49 years old) with a recent birth (<2 years) reporting postnatal care by any provider for within 2 days (0-48 hours) after her most recent delivery.
Proportion of women receiving antenatal care 4 or more times during pregnancy | Change between pre (baseline) and post (endline-up to 36 months) intervention
  Percentage of women (15-49 years old) reporting four or more antenatal care visits at a health facility during their most pregnancy, where their last pregnancy was completed within two years of survey

CONTACTS AND LOCATIONS:
Overall Officials: Dismas K Matovelo, MD, MMed, Principal Investigator — Catholic University of Health and Allied Sciences
Locations (1):
- Catholic University of Health and Allied Sciences, Mwanza, Tanzania

IPD SHARING:
Plan to Share IPD: Yes
De-Identified data will be shared with district officials, government offices and other stakeholders

REFERENCES:
- [Derived] Matovelo D, Boniphace M, Singhal N, Nettel-Aguirre A, Kabakyenga J, Turyakira E, Mercader HFG, Khan S, Shaban G, Kyomuhangi T, Hobbs AJ, Manalili K, Subi L, Hatfield J, Ngallaba S, Brenner JL. Evaluation of a comprehensive maternal newborn health intervention in rural Tanzania: single-arm pre-post coverage survey results. Glob Health Action. 2022 Dec 31;15(1):2137281. doi: 10.1080/16549716.2022.2137281. PMID 36369729
- See also: Mama na Mtoto website — https://www.mnmtanzania.com/